CLINICAL TRIAL: NCT03790345
Title: Effect of Vitamin B6 and B12 in the Treatment of Movement Disorders Induced by Antipsychotics
Brief Title: Vitamin B6 and B12 in the Treatment of Movement Disorders Induced by Antipsychotics
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B12B16study
Record Dates: First submitted 2018-12-21; First posted 2018-12-31 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2018-12

CONDITIONS: Schizophrenia; Drug Induced Movement Disorder, Unspecified; Oxidative Stress
Keywords: Schizophrenia; Cobalamin; Pyridoxine; Drug-induced movement disorder
MeSH Terms: conditions — Schizophrenia | interventions — Pyridoxine; Vitamin B 6; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: Proof of concept 12-week prospective, randomized, double-blind, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): 15 subjects will be randomly assigned to adjuvant treatment with 200mg of vitamin B6 (pyridoxine).
  Interventions: Drug: Pyridoxine
- Experimental group 2 (Experimental): 15 subjects will be randomly assigned to adjuvant treatment with 2mg of vitamin B12 (cobalamin).
  Interventions: Drug: Cobalamin
- Placebo oral tablet (Sham Comparator): 15 subjects will be randomly assigned to adjuvant treatment with placebo.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Pyridoxine — Adjuvant daily treatment with 200mg of pyridoxine
  Other Names: Vitamin B6
  Arms: Experimental group 1
Drug: Cobalamin — Adjuvant daily treatment with 2mg of cobalamin
  Other Names: Vitamin B12
  Arms: Experimental group 2
Drug: Placebo Oral Tablet — Adjuvant daily treatment with placebo
  Arms: Placebo oral tablet

SUMMARY:
D2 dopaminergic receptor blockers, used to treat schizophrenia, can lead to the onset of movement disorders. Drug-induced movement disorders encompass several syndromes. Parkinsonism, dystonia, dyskinesia and akathisia are the most prevalent. All of them lead to poor adherence to the treatment instituted, decrease in the quality of life, relapses and hospitalizations. The pathophysiology of drug-induced movement disorders is complex and poorly understood, but seems to be associated with oxidative stress, as a result of an increase in free radicals generated from dopamine metabolism. Treatment strategies following the onset of drug-induced movement disorders include neuroleptic discontinuation, use of atypical antipsychotics and anticholinergics. A pre-clinical study showed that the antioxidant properties of vitamins B6 and B12, alone or in combination, prevented the development of orofacial dyskinesia induced by haloperidol. This clinical trial aims to evaluate the effects of vitamins B6 and B12 on the treatment of patients diagnosed with schizophrenia, schizoaffective or bipolar disorder who present with tardive dyskinesia, dystonia and parkinsonism.

DETAILED DESCRIPTION:
D2 dopaminergic receptor blockers, used to treat schizophrenia, can lead to the onset of drug-induced movement disorders, such as parkinsonism, dystonia, dyskinesia and akathisia. They seem to be associated with oxidative stress, as a result of an increase in free radicals generated from dopamine metabolism. A preclinical study showed that vitamin B6 (pyridoxine) and B12 (cobalamin), alone or in combination, prevented the development of orofacial dyskinesia induced by haloperidol in an animal model of schizophrenia.

Specific Aim1: To conduct a prospective, randomized, double-blind, placebo-controlled trial to evaluate the efficacy of 12-week adjuvant treatment with 200mg of pyridoxine (B6) or 2mg of cobalamin (B12) to treat drug-induced movement disorders of patients with schizophrenia, schizoaffective or bipolar disorder. The investigators will randomly assign 45 patients into three groups: placebo, B6 or B12 and check whether administration of vitamin B6 (pyridoxine) or B12 (cobalamin) attenuates drug-induced movement disorders (IDDM) in patients with diagnosis of schizophrenia, schizoaffective or bipolar disorder.

Specific Aim 2: To quantify changes in serum markers of inflammation and biomarkers of oxidative stress in response to adjunctive treatment with B6 or B12. The hypothesis is that changes in these biomarkers will mediate the clinical response to them.

Research Plan: The investigators will carry out a proof of concept 12-week prospective, randomized, double-blind, controlled trial of vitamin B6 and B12, at doses of 200 mg/day and 2mg/day, respectively, or identical placebo tablets, added to ongoing antipsychotics in 45 stable patients (ages 18-60 years, 15 patients per group) with diagnosis of schizophrenia, schizoaffective or bipolar disorder. The study will be conducted at the Drug Research and Development Center (NPDM), at the Universidade Federal do Ceará, Fortaleza, Brazil. This center has a long history of performing placebocontrolled trials in clinical medicine (http://www.npdm.ufc.br/) and has the necessary infrastructure to successfully complete the proposed study protocol. All participants will give written informed consent prior to study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent;
* Schizophrenia diagnosis (confirmed by Structured Clinical Interview (SCID);
* Movement disorders induced by psychotropic drugs of at least moderate severity;
* Exposure to psychotropic medication for at least three months prior of the appearance of movement disorders;.
* Disorders of movement for at least one year;
* Stable psychotropic regimen for at least one month prior to study entry.

Exclusion Criteria:

* 6-month history of any drug or alcohol abuse or dependence;
* Changes in psychotropic medications within the last 4 weeks;
* General medical illness including autoimmune disorders, known chronic infections such as HIV or hepatitis C, and liver or renal failure that could adversely impact on patient outcome;
* Women who are planning to become pregnant, are pregnant, or are breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-06-03 (Estimated); Study Completion 2021-11-03 (Estimated)

PRIMARY OUTCOMES:
Change in the Simpson-Angus Extrapyramidal Symptoms Scale (SAS) scores | Baseline and 12 weeks
  10-item rating scale to assess extrapyramidal symptoms; each item is scored 0-4, yielding a total between 0 and 40.
Change in the Barnes Akathisia Rating Scale (BAS, BARS) scores | Baseline and 12 weeks
  Objective Akathisia, Subjective Awareness of Restlessness and Subjective Distress Related to Restlessness are rated on a 4-point scale from 0 - 3 and are summed yielding a total score ranging from 0 to 9. The Global Clinical Assessment of Akathisia uses a 5-point scale ranging from 0 - 4.
Change in the Abnormal Involuntary Movement Scale (AIMS) scores | Baseline and 12 weeks
  10-item rating scale to assess involuntary movements; items are rated on a five-point scale of severity from 0-4, yielding a total between 0 and 40.

SECONDARY OUTCOMES:
Change in the Brief Psychiatry Rating Scale (BPRS) scores | Baseline and 12 weeks
  18-item rating scale to assess changes in psychopathology; each item is scored 0-6, yielding a total between 0 and 40.
Change in Plasma Glutathione (GSH) | Baseline and 12 weeks
  GSH in ng/mL
Change in serum level of Nitrite | Baseline and 12 weeks
  Nitrite in nanomole/mililiter
Change in serum level of Thiobarbituric acid reactive substances (TBARS) | Baseline and 12 weeks
  TBARS in mmol of malonaldehyde/mL
Change in serum level of Interleukin 1 β (IL-1β) | Baseline and 12 weeks
  IL-1β in pg/mL
Change in serum level of Interleukin-4 | Baseline and 12 weeks
  IL-4 in pg/mL
Change in serum level of Interferon gamma (IFNγ) | Baseline and 12 weeks
  IFNγ in pg/mL
Change in serum level of Tumor necrosis factor alpha (TNF-α) | Baseline and 12 weeks
  TNF-α in pg/mL
Change in Indoleamine 2,3-dioxygenase (IDO) enzymatic activity | Baseline and 12 weeks
  IDO activity in U IDO mol^-1/mg^-1

CONTACTS AND LOCATIONS:
Overall Officials: Lia LO Sanders, MD, PhD, Principal Investigator — Núcleo de Pesquisa e Desenvolvimento de Medicamentos
Locations (1):
- Núcleo de Pesquisa e Desenvolvimento de Medicamentos - UFC, Fortaleza, Ceará, Brazil